CLINICAL TRIAL: NCT05704868
Title: UniVRse: Pilot Randomised Controlled Trial of Virtual Reality Cognitive Behaviour Therapy (VR-CBT) for Students With Social Anxiety
Brief Title: UniVRse: VR-CBT for Students With Social Anxiety
Acronym: UniVRse
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: University of Westminster (Other); University of Nottingham (Other); University of Sussex (Other)
Responsible Party: Principal Investigator, Cassie Hazell, Lecturer B, University of Surrey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETH2122-3503
Record Dates: First submitted 2022-12-12; First posted 2023-01-30 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Social Anxiety
Keywords: Social anxiety; Students; University; Virtual Reality; Cognitive Behaviour Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UniVRse + TAU (Experimental): UniVRse is a Virtual Reality (VR) intervention targeting social anxiety in students using cognitive behavioural therapy (CBT) techniques - specifically graded exposure. Participants will have access to UniVRse for a month post-randomisation and it is recommended they complete 6 sessions each 30-minutes long over this period. Exposure to the intervention will be reached if participants complete 2 30-minute sessions. UniVRse is a self-help intervention meaning that participants can engage in the intervention independently. Participants will be supported to progress through the UniVRse programme by a virtual mentor called Sam that will take on the role traditionally undertaken by the 'therapist'. Sam's function will be to provide psychoeducation, provide instruction on how to use the VR kit and interact with the virtual environment, and provide support and encouragement. Participants will be able to complete the intervention either on campus or at home.
  Interventions: Behavioral: UniVRse + TAU
- Waitlist + TAU (No Intervention): We will be using a wait list control group. The wait list control group will receive treatment as usual for the duration of the trial. Treatment as usual may include active monitoring, meetings with academic advisors, psychiatric medication, and/or support from an NHS mental health team. We will not withhold treatment from the control group, but prospective participants may not be eligible to take part if they have current or confirmed plans to receive a psychology therapy (see exclusion criteria). Once the trial has ended, the participants in the control arm will be the first to be offered UniVRse when it is taken up by university support services.

INTERVENTIONS:
Behavioral: UniVRse + TAU — UniVRse uses well-established evidence-basedcognitive behavioural therapy (CBT) techniques - specifically graded exposure - to reduce fear and worries about social situations. People work towards overcoming their anxiety in a step-by-step fashion, building up to the most feared situation. In the context of UniVRse, students will be presented with four university-based scenarios that our coproduction team identified as being the most anxiety-induing for students:
  1. Attending a lecture;
  2. Group work in a seminar;
  3. Delivering a presentation;
  4. Contributing to an online seminar.
  The UniVRse programme has been designed with our co-production team comprised of tirst-generation students with social anxiety, CBT therapists, and a VR design company.
  Arms: UniVRse + TAU

SUMMARY:
The goal of this pilot randomised controlled trial is to evaluate the effectiveness of the UniVRse VR-CBT programme in students with social anxiety. The aims of this trial are:

1. To determine whether a full trial is justified;
2. To establish the effect size on the co-primary outcomes for a sample size calculation for a definitive trial;
3. To address questions concerning study recruitment, retention, and acceptability.

Participants will complete a baseline assessment (T0) and then be randomly allocated to receive either UniVRse VR-CBT or join the wait-list control group. UniVRse VR-CBT uses graded exposure techniques delivered using VR to help students feel more confident in university-based situations. Data will be collected post-intervention (T1) along with exit interviews to assess participant experience.

ELIGIBILITY:
Inclusion Criteria:

For participants to be eligible to take part, they must be:

* A current student at the University of Westminster;
* Able to read and communicate in English;
* Wanting help to feel more confident at university;
* Deemed to have context-specific social anxiety as defined by a response of 'moderate' or 'often' on one of the subscales from any one of the following items from the MLSAS-SR: 5, 12, 17, and 9. These items reflect the highest level (i.e. most anxiety-invoking) of each of the four scenarios within the UniVRse programme:

  * Asking a question in a lecture in person
  * Delivering a presentation on your own in front of the class
  * Speaking using my mic during online seminars
  * Speaking up during small group discussions in person

Exclusion Criteria:

Persons will be excluded from the study if meet any of the following criteria:

* Have photosensitive epilepsy;
* Have a visual impairment that cannot be corrected with glasses;
* Have a balance disorder;
* Have a significant auditory impairment;
* Have current and active suicidal plans;
* Are currently accessing or have confirmed plans to access another psychological intervention during the course of the study.

Participants will be excluded from providing a saliva sample (required for the cortisol measurement) if they meet any of the following criteria:

* Are pregnant;
* Currently breastfeeding;
* Taking any medications;
* Have any other serious medical condition;
* Think that they currently have COVID-19. These participants may still participate in the wider UniVRse trial if they meet all of the aforementioned main trial inclusion/exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Social Phobia Inventory (SPIN) | One week
  The Social Phobia Inventory (SPIN) (Connor et al., 2000) is a 17-item questionnaire measuring social anxiety.
Modified Liebowitz Social Anxiety Scale (MLSAS-SR) | One week
  We have used the LSAS-SR as the basis for developing a social anxiety scale that is specific to the university environment. The modified version of this scale has a list of different university-based situations and participants are asked the extent to which they fear and avoid each of the situations.

SECONDARY OUTCOMES:
Patient Health Questionnaire 9 (PHQ-9) | Last 2 weeks
  The PHQ-9 (Spitzer et al., 1999) measures levels of depression.
Generalised Anxiety Disorder 7 (GAD-7) | Last 2 weeks
  Developed by the same research team as the PHQ-9, the GAD-7 (Spitzer et al., 2006) is a brief screening tool used in primary care to assess the severity of generalised anxiety symptoms.
The Rathus Assertiveness Schedule (RAS) | One day
  The RAS (Rathus, 1973) was developed to measure general assertiveness.
Spreitzer's Psychological Empowerment Scale (SPES) | One week
  The SPES (Spreitzer, 1995) assesses assertiveness in a specific context in terms of feeling empowered.
Short Instrument for measuring students' Confidence with Key Skills (SICKS) | One week
  The SICKS (Bray et al., 2020) assesses students' confidence in relation to a range of education-related activities.
Rosenberg self-esteem scale (RSES) | One day
  The RSES (Rosenberg, 1965) assesses global self-esteem.
Question of Belonging (QoB) | One week
  The QoB (Walton & Cohen, 2007) assesses the extent to which students feel like they belong within their university community.
Identification with University (IwU) | One week
  The IwU (Nieuwenhuis et al., 2019) is a subscale within a broader assessment on social identity. The IwU assesses the extent to which persons perceive being a university student is consistent with their social identity.
Domain Specific Hope Scale - Social Hope (DSHS-SH) and Academic Hope (DSHS-AH) subscales | One day
  The DSHS assesses hope in relation to a variety of life domains. There are a total of six subscales and in this study we will be utilising both the social and academic hope subscales (Sympson, 1999).
Attendance | Two weeks
  The University of Westminster has a 'tap in' system whereby students are required to use their student ID to register their attendance for all timetabled activities. These data are used to assess student attendance and identify any students at risk of disengaging.
Cortisol in saliva samples | Three days
  We will ask participants to provide 6 saliva samples a day for three consecutive days per time point i.e., 6 each at T0 on days 1, 2, and 3, and 6 each at T1 on days 1, 2, and 3 - this equates to 18 saliva samples her time point and 36 samples in total across the duration of the study per participant. We will use the samples to measure levels of the stress hormone cortisol.

OTHER OUTCOMES:
Edinburgh adverse effects of psychological therapy (EDAPT) | One month
  The EDAPT (Mc Glanaghy et al., 2021) was developed via a Delphi consultation with experts by experience and profession. The EDAPT is a checklist of 42 items each reflecting a potential adverse event that could occur after receiving a psychological therapy.
IAPT Patient Experience Questionnaire (IAPT-PEQ) | One month
  To assess how participants experienced the intervention, we will adapt the PEQ used in IAPT services (Clarke, 2011).
Friends and family test (FFT) | One month
  The FFT (Department of Health, 2013) is used across all NHS services as a measure of patient satisfaction.
Simulator Sickness Questionnaire (SSQ) | One month
  The SSQ (Kennedy et al., 1993) measures the presence of potential negative effects associated with using VR.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Westminster, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hazell CM, Malinowski J, Edwards B, Bergin ADG, Berry C, Flynn M, Smyth N, Birkett J. UniVRse: protocol for a pilot randomised controlled trial of virtual reality cognitive-behaviour therapy for students with social anxiety. Pilot Feasibility Stud. 2026 Feb 5. doi: 10.1186/s40814-026-01771-4. Online ahead of print. PMID 41645300
- See also: Project website — http://blog.westminster.ac.uk/univrse/